CLINICAL TRIAL: NCT06564064
Title: The Effect of Abdominal Binders on Patient's Wellbeing After Cesarean Delivery :a Prospective Comparative Study
Brief Title: The Effect of Abdominal Binders on Patient's Wellbeing After Cesarean Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Saad Abdellattif, Sohag - El Maragha city, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-24-07-20MS
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Effect of Abdominal Binders on Patient ( Pain, Quality of Recovery ) After Cesaean Section
Keywords: binders, cesarean section , VAS, QOR 40
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: study group (abdominal binders) and control group
Who Masked: Participant, Investigator
Masking Description: participant and investigator both are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group Study group(Group1) (Active Comparator): 25 participant will be in study group (abdominal binders)
  Interventions: Device: abdominal binder
- Control group (Group 2) (Placebo Comparator): 25 participants will be in control group
  Interventions: Device: abdominal binder

INTERVENTIONS:
Device: abdominal binder — study group will be abdominal binders and control group will be control group , 12 hrs and one week later VAS and QOR 40 will assess patient,s wellbeing

SUMMARY:
The effect of abdominal binders on patient's wellbeing after cesarean delivery

DETAILED DESCRIPTION:
The effect of abdominal binders on patient's wellbeing after cesarean delivery 12 hours and one week after cesarean section

ELIGIBILITY:
Inclusion Criteria:

any female post cesarean section of singleton 34 wks gestaion fetus with previous cs

Exclusion Criteria:

primary cs any hypertensive disorder with pregnancy any neurologiacal disease general anasthesia or vertical incision

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female
Enrollment: 50 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
The effect of abdominal binders on pain after cesarean section | 6 months
  abdominal binders will be fit on patient abdomin 2 hrs post cs and VAS will be assessed 12 hrs post cesarean section

SECONDARY OUTCOMES:
The effect of abdominal binders on patient's wellbeing after cesarean delivery | one week postoperatively
  effect after one week on quality of recovery ( infection, hematoma, seroma) by QOR 40

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Ghana S, Hakimi S, Mirghafourvand M, Abbasalizadeh F, Behnampour N. Randomized controlled trial of abdominal binders for postoperative pain, distress, and blood loss after cesarean delivery. Int J Gynaecol Obstet. 2017 Jun;137(3):271-276. doi: 10.1002/ijgo.12134. Epub 2017 Mar 28. PMID 28241386
- [Background] Gustafson JL, Dong F, Duong J, Kuhlmann ZC. Elastic Abdominal Binders Reduce Cesarean Pain Postoperatively: A Randomized Controlled Pilot Trial. Kans J Med. 2018 May 18;11(2):1-19. eCollection 2018 May. PMID 29796155
- [Background] Karaca I, Ozturk M, Alay I, Ince O, Karaca SY, Erdogan VS, Ekin M. Influence of Abdominal Binder Usage after Cesarean Delivery on Postoperative Mobilization, Pain and Distress: A Randomized Controlled Trial. Eurasian J Med. 2019 Oct;51(3):214-218. doi: 10.5152/eurasianjmed.2019.18457. PMID 31692751
- [Background] Saeed S, Rage KA, Memon AS, Kazi S, Samo KA, Shahid S, Ali A. Use of Abdominal Binders after a Major Abdominal Surgery: A Randomized Controlled Trial. Cureus. 2019 Oct 3;11(10):e5832. doi: 10.7759/cureus.5832. PMID 31754567
- [Background] Terkawi AS, Tsang S, Abolkhair A, Alsharif M, Alswiti M, Alsadoun A, AlZoraigi US, Aldhahri SF, Al-Zhahrani T, Altirkawi KA. Development and validation of Arabic version of the Short-Form McGill Pain Questionnaire. Saudi J Anaesth. 2017 May;11(Suppl 1):S2-S10. doi: 10.4103/sja.SJA_42_17. PMID 28615999
- [Background] Terkawi AS, Myles PS, Riad W, Nassar SN, Mahmoud M, AlKahtani GJ, Sala FJ, Abdulrahman A, Doais KS, Terkawi RS, Tsang S. Development and validation of Arabic version of the postoperative quality of recovery-40 questionnaire. Saudi J Anaesth. 2017 May;11(Suppl 1):S40-S52. doi: 10.4103/sja.SJA_77_17. PMID 28616003